CLINICAL TRIAL: NCT01780675
Title: Prophylactic Cranial Irradiation With or Without Hippocampal Avoidance in SCLC a Randomized Phase III Trial
Brief Title: Hippocampus Avoidance PCI vs PCI
Acronym: HA-PCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M12PHA
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Small Cell Lung Cancer; Lung Cancer
Keywords: Prophylactic Cranial Irradiation; Hippocampal Avoidance Prophylactic Cranial Irradiation
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic Cranial Irradiation (Active Comparator): Radiation. Prophylactic Cranial Irradiation: 10 times 2.5 Gy (total 25 Gy)
  Interventions: Radiation: Radiation Prophylactic Cranial Irradiation
- Hippocampal Avoidance PCI (Experimental): Radiation. Hippocampal Avoidance PCI. 10 times 2.5 Gy (total 25 Gy).
  Interventions: Radiation: Radiation Hippocampal Avoidance PCI

INTERVENTIONS:
Radiation: Radiation Prophylactic Cranial Irradiation
  Arms: Prophylactic Cranial Irradiation
Radiation: Radiation Hippocampal Avoidance PCI
  Arms: Hippocampal Avoidance PCI

SUMMARY:
Using Intensity Modulated radiotherapy it is possible to treat the entire brain to standard dosages of whole-brain radiation, while keeping the radiation dose to the hippocampus low. However, a clear relationship between radiation dose and damage to the hippocampal stem cells has not been established yet.

This study is initiated to investigate the early and delayed neurotoxicity of PCI and to assess in a randomised design the benefits and risks of sparing the hippocampus in Small Cell Lung Cancer patients who receive PCI.

ELIGIBILITY:
Inclusion Criteria:

* - Small Cell Lung Cancer patients (stage I-III or stage IV without clinical or radiological evidence of brain metastases) candidate for PCI, i.e. without progressive disease after chemo-radiotherapy in stage I-III or after a remission after chemotherapy in stage IV
* Sufficient proficiency in Dutch

Exclusion Criteria:

* Prior radiotherapy to the brain
* Clinical evidence for brain metastases or primary brain tumors- Evidence of progressive extracranial metastatic disease
* Previous malignancy < 2 years ago except for adequately treated basal cell carcinoma of the skin and carcinoma in situ of the cervix
* Any systemic anticancer treatment during PCI or within 3 weeks before start PCI
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-04; Primary Completion 2019-04-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
neurocognitive decline | 4 months
  Each patient's total recall score recorded at 4 months will be compared to baseline and dichotomized into success (decline less or equal 5 points) or failure (decline more than 5 points). The difference between the groups, in terms of dichotomized decline will be tested by means of the Fisher's exact test. A p-value less than 0.049 will be considered significant. The primary analysis will be based on an intention-to-treat principle.

SECONDARY OUTCOMES:
safety | 2 years
  Brain metastases Time from randomization to the occurrence of brain metastases will be calculated and depicted in a cumulative incidence plot. Sensitivity analysis will be performed to assess the value of PCI vs HA-PCI treatment once considering patients dying without distant brain metastases to be censored and once using competing risk analysis considering distant metastases and death as separate events

CONTACTS AND LOCATIONS:
Overall Officials: Jose Belderbos, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (9):
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Netherlands (6):
  - The Netherlands Cancer Institute, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC Cancer Centre, Rotterdam
  - Instituut Verbeeten, Tilburg

REFERENCES:
- [Derived] Zeng H, Schagen SB, Hendriks LEL, Sanchez-Benavides G, Jaspers JPM, Manero RM, Lievens Y, Murcia-Mejia M, Kuenen M, Rico-Oses M, Albers EAC, Samper P, Houben R, de Ruiter MB, Dieleman EMT, Lopez-Guerra JL, De Jaeger K, Counago F, Lambrecht M, Calvo-Crespo P, Belderbos JSA, De Ruysscher DKM, Rodriguez de Dios N. Impact of HA-PCI on self-reported cognitive functioning and brain metastases in small-cell lung cancer: Pooled findings of NCT01780675 and PREMER trials. Lung Cancer. 2025 Jan;199:108036. doi: 10.1016/j.lungcan.2024.108036. Epub 2024 Nov 23. PMID 39615412
- [Derived] Ishibashi A, Kurosaki H, Miura K, Utsumi N, Sakurai H. Influence of Modulation Factor on Treatment Plan Quality and Irradiation Time in Hippocampus-Sparing Whole-Brain Radiotherapy Using Tomotherapy. Technol Cancer Res Treat. 2021 Jan-Dec;20:15330338211045497. doi: 10.1177/15330338211045497. PMID 34632876